CLINICAL TRIAL: NCT06089135
Title: Shockwave Lithoplasty Compared to Cutting Balloon Treatment in Calcified Coronary Disease - A Randomized Controlled Trial (Short-Cut)
Brief Title: Shockwave Lithoplasty Compared to Cutting Balloon Treatment in Calcified Coronary Disease - A Randomized Controlled Trial
Acronym: Short-Cut
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baim Institute for Clinical Research (Other)
Collaborators: Robert W. Yeh, MD (Unknown); Ajay Kirtane, MD (Unknown); C. Michael Gibson, MS, MD (Unknown); Kathleen Kearney, MD (Unknown); Akiko Maehara, MD (Unknown); Suzanne Baron, MD (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BBC22
Record Dates: First submitted 2023-10-06; First posted 2023-10-18 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Treatment in Calcified Coronary Disease
Keywords: Intravascular Lithoplasty; Cutting Balloon; Calcified Coronary Disease; Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intravascular Lithotripsy (Active Comparator)
  Interventions: Device: Intravascular Lithotripsy
- Cutting Balloon (Active Comparator)
  Interventions: Device: Cutting Balloon

INTERVENTIONS:
Device: Intravascular Lithotripsy — Intravascular lithotripsy will be performed with or without rotational atherectomy prior to drug-eluting stent implantation in patients with moderate to severely calcified coronary arteries.
  Arms: Intravascular Lithotripsy
Device: Cutting Balloon — Cutting Balloon therapy will be performed with or without rotational atherectomy prior to drug-eluting stent implantation in patients with moderate to severely calcified coronary arteries.
  Arms: Cutting Balloon

SUMMARY:
The Short-Cut trial is a prospective, investigator-initiated, multicenter, randomized controlled trial that is designed to compare the efficacy of cutting balloon angioplasty vs. intravascular lithotripsy prior to drug-eluting stent implantation in patients with moderate to severely calcified coronary arteries.

DETAILED DESCRIPTION:
The trial will be composed of two cohorts:

* Patients treated with up-front rotational atherectomy
* Patients in whom atherectomy is not planned

Randomization to either cutting balloon angioplasty or intravascular lithotripsy will occur as follows in the 2 cohorts:

* After rotational atherectomy is safely completed In the rotational atherectomy arm
* After safe and successful wire crossing in patients in whom atherectomy is not planned.

The trial is designed to demonstrate non-inferiority between cutting balloon angioplasty and intravascular lithotripsy in each cohort with regards to the primary endpoint of post-procedural stent area as measured by intravascular imaging at the site of maximal calcification.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subject is > 21 years old 2. Subject with an indication for PCI for the treatment of a) stable coronary artery disease; b) unstable angina; or c) NSTEMI with evidence of down-trending biomarkers 3. Subject is willing and able to provide informed written consent Angiographic Inclusion Criteria

  1. The target lesion is a de novo native coronary lesion
  2. The target vessel is a native coronary artery with either:

     1. A stenosis > 70%; or,
     2. A stenosis > 50% and <70% with evidence of ischemia via either positive stress test, FFR value < 0.80 or RFR/iFR/DFR value < 0.89
  3. The reference diameter of the target vessel is > 2.5mm and < 4.0 mm at the lesion site
  4. The target lesion has evidence of significant calcium at the lesion site defined either as,

     1. The presence of radiopacities involving both sides of the arterial wall > 5mm and involving the target lesion on angiography
     2. the presence of > 270o arc of superficial calcium on intravascular imaging with a length > 5mm or the presence of 360o arc of superficial calcium

        Exclusion Criteria:

  <!-- -->

  1. Patient is pregnant
  2. Patient is actively participating in another clinical trial
  3. Known LVEF < 25%
  4. Ongoing Non-STEMI with rising biomarkers
  5. Cardiogenic shock or requirement for mechanical/pharmacologic hemodynamic support
  6. Planned use in the randomized lesion of a bare metal stent or non-stent treatment only
  7. Patient has a known allergy to contrast which cannot be adequately pre-treated
  8. Patient has a history of bleeding or coagulopathy and is unable to receive blood transfusion if needed
  9. Patient presents with STEMI
  10. Patient is unable to tolerate dual anti-platelet therapy
  11. Patient has suffered a recent cerebrovascular event (stroke/TIA) within last 30 days

      Angiographic Exclusion Criteria

  <!-- -->

  1. Presence of large thrombus in the target vessel
  2. Inability to pass coronary guidewire across the lesion
  3. The target vessel has excessive tortuosity (Defined as presence of 2+ bends > 90o or 3+ bends > 75o) or other anatomic considerations that precludes intravascular imaging
  4. The target lesion is within a coronary artery bypass graft
  5. The target lesion involves a bifurcation lesion in which either a 2-stent strategy is planned or both branches are planned for calcium modification
  6. Coronary artery disease that requires surgical revascularization
  7. Angiographic or imaging evidence of dissection in the target vessel prior to randomization
  8. Investigator feels there is not equipoise regarding the treatment strategy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 2023-12-31 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Primary Endpoint | 30 days
  Post-procedural stent area at the point of maximum calcification as measured by intravascular imaging

SECONDARY OUTCOMES:
Procedural Cost | Index procedure
Procedural success | Index procedure
  Procedural success defined as stent delivery with a residual stenosis < 20% in the absence of significant angiographic complication (e.g. severe dissection, perforation, abrupt closure or no-reflow) with final TIMI 3 flow in the target vessel and the absence of intra-procedural death
Angiographic success | Index procedure
  Angiographic success defined as stent delivery with a residual stenosis < 20% in the absence of significant angiographic complication (e.g. severe dissection, perforation, abrupt closure or no-reflow)
Strategy success | Index procedure
  Strategy success defined as stent delivery with a residual stenosis < 20% in the absence of significant angiographic complication (e.g., severe dissection, perforation, abrupt closure or no-reflow and not having to use an alternative calcium modification device (e.g. atherectomy device or specialty balloon other than routine non-compliant balloon)
Peri-procedural Myocardial Infarction | within 48 hours of index procedure
  Peri-procedural Myocardial Infarction as defined by Academic Research Consortium-2
In-hospital MACCE | hospitalization
  In-hospital MACCE defined as composite of all-cause death, unplanned urgent target vessel revascularization, unplanned cardiothoracic surgery, spontaneous myocardial infarction or stroke/TIA at hospital discharge.
30 Day MACCE | 30 days
  30 Day MACCE defined as composite of all-cause death, unplanned target vessel revascularization, unplanned cardiothoracic surgery, spontaneous myocardial infarction or stroke/TIA at 30 days

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - UAB Structural Heart and Valve Clinic, Birmingham, Alabama
  - Banner Health, Phoenix, Arizona
  - Honor Health, Scottsdale, Arizona
  - UCSF Cardiology, San Francisco, California
  - Yale School of Medicine, New Haven, Connecticut
  - Saint Luke's, Overland Park, Kansas
  - Maine Medical Center, Portland, Maine
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medcial Center, Boston, Massachusetts
  - Henry Ford Health, Detroit, Michigan
  - Capital Cardiology, Albany, New York
  - Columbia Cardiology, New York, New York
  - Columbia University Medical Center/ NewYork Presbyterian Hospital, New York, New York
  - Christ Hospital, Cincinnati, Ohio
  - UPMC, Pittsburgh, Pennsylvania
  - Wellspan York Hospital, York, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Heart and Vascular Hospital, Dallas, Texas
  - Houston Methodist, Houston, Texas
  - Baylor Scott and White Health, Plano, Texas
  - UVA Heart and Vascular Center, Charlottesville, Virginia
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shah M, Najam O, Bhindi R, De Silva K. Calcium Modification Techniques in Complex Percutaneous Coronary Intervention. Circ Cardiovasc Interv. 2021 May;14(5):e009870. doi: 10.1161/CIRCINTERVENTIONS.120.009870. Epub 2021 Jan 14. PMID 33441017
- [Background] Allali A, Toelg R, Abdel-Wahab M, Hemetsberger R, Kastrati A, Mankerious N, Traboulsi H, Elbasha K, Rheude T, Landt M, Geist V, Richardt G. Combined rotational atherectomy and cutting balloon angioplasty prior to drug-eluting stent implantation in severely calcified coronary lesions: The PREPARE-CALC-COMBO study. Catheter Cardiovasc Interv. 2022 Nov;100(6):979-989. doi: 10.1002/ccd.30423. Epub 2022 Oct 19. PMID 36262074
- [Background] Furuichi S, Tobaru T, Asano R, Watanabe Y, Takamisawa I, Seki A, Sumiyoshi T, Tomoike H. Rotational atherectomy followed by cutting-balloon plaque modification for drug-eluting stent implantation in calcified coronary lesions. J Invasive Cardiol. 2012 May;24(5):191-5. PMID 22562910
- [Background] Abdel-Wahab M, Toelg R, Byrne RA, Geist V, El-Mawardy M, Allali A, Rheude T, Robinson DR, Abdelghani M, Sulimov DS, Kastrati A, Richardt G. High-Speed Rotational Atherectomy Versus Modified Balloons Prior to Drug-Eluting Stent Implantation in Severely Calcified Coronary Lesions. Circ Cardiovasc Interv. 2018 Oct;11(10):e007415. doi: 10.1161/CIRCINTERVENTIONS.118.007415. PMID 30354632
- [Background] Mangieri A, Nerla R, Castriota F, Reimers B, Regazzoli D, Leone PP, Gasparini GL, Khokhar AA, Laricchia A, Giannini F, Casale F, Bezzeccheri A, Briguori C, Colombo A. Cutting balloon to optimize predilation for stent implantation: The COPS randomized trial. Catheter Cardiovasc Interv. 2023 Mar;101(4):798-805. doi: 10.1002/ccd.30603. Epub 2023 Feb 25. PMID 36841945
- [Background] Kereiakes DJ, Hill JM, Shlofmitz RA, Klein AJ, Riley RF, Price MJ, Herrmann HC, Bachinsky W, Waksman R, Stone GW; Disrupt CAD III Investigators. Intravascular Lithotripsy for Treatment of Severely Calcified Coronary Arteries: 2-Year Results-Disrupt CAD III Study. JACC Cardiovasc Interv. 2023 Oct 9;16(19):2472-2474. doi: 10.1016/j.jcin.2023.07.010. Epub 2023 Sep 6. No abstract available. PMID 37676225